CLINICAL TRIAL: NCT02197416
Title: Open Label, Single Arm Safety Prospective Cohort Study of Dabigatran Etexilate for Secondary Prevention of Venous Thromboembolism in Children From 0 to Less Than 18 Years
Brief Title: Safety of Dabigatran Etexilate in Blood Clot Prevention in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1160.108; 2014-000583-18 (EudraCT Number)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Venous Thromboembolism; Secondary Prevention
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- dabigatran etexilate (Experimental)
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — Age and weight appropriate capsule dose (combination of 50 mg, 75 mg and 110 mg capsules) or pellets or oral liquid formulation

SUMMARY:
This open-label, single arm prospective cohort study will assess the safety of dabigatran etexilate in secondary prevention of venous thromboembolism in paediatric patients. Children from 0 to less than 18 years of age will be eligible to participate.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects 0 to less than 18 years of age at the time of informed consent / assent
* Previously documented objective diagnosis of VTE, followed by completed course of initial VTE treatment for at least 3 months (in case of VKA - intended INR between 2 and 3) or completed study treatment (i.e. reached Visit 8) in the 1160.106 trial. Patients, who during the treatment phase of 1160.106 trial were switched from dabigatran etexilate to SOC arm for any reason, are not eligible for this study.
* Presence of an unresolved clinical risk factor requiring further anticoagulation for secondary VTE prevention (e.g. central venous line, underlying disease, thrombophilia, etc.)
* Written informed consent form (ICF) provided by the patient's parent or legal guardian and assent provided by the patient (if applicable) at the time of ICF signature according to local regulations.
* Further inclusion criteria apply

Exclusion criteria:

* Conditions associated with an increased risk of bleeding
* Renal dysfunction (eGFR < 50 mL/min/1.73m^2 using the Schwartz formula) or requirement for dialysis. eGFR retesting during the screening period is allowed (once).
* Active infective endocarditis
* Subjects with a heart valve prosthesis requiring anticoagulation.
* Hepatic disease: Active liver disease, including known active hepatitis A, B or C or Persistent alanine aminotransferase (ALT) or aspartate transaminase (AST) or alkaline phosphatase (AP) > 3 × upper limit of normal (ULN) within 3 months of screening
* Pregnant or breast feeding females. Females who have reached menarche and are not using an acceptable method of birth control, or do not plan to continue using this method throughout the study and / or do not agree to adhere to pregnancy testing required by this protocol
* Patients in age group 0 to < 2 years with gestational age at birth < 37 weeks or with body weight lower than the 3rd percentile
* Anemia (hemoglobin < 80g/L) or thrombocytopenia (platelet count < 80 x 109/L) at screening. Transfusions during the screening period are allowed, provided that a satisfactory hemoglobin or platelet level is attained prior to visit 2
* Patients who have taken restricted medication prior to first dose of study medication
* Patients who have received an investigational drug in the past 30 days prior to screening, except patients who have completed the treatment period (up to Visit 8) in 1160.106 trial
* Patients who are allergic/sensitive to any component of the study medication including solvent
* Patients or parents/legal guardians considered unreliable to participate in the trial per investigator judgment or any condition which would present a safety hazard to the patient based on investigator judgment
* Further exclusion criteria apply

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (62):
- United States (9):
  - University of California Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Alliance for Childhood Diseases, Las Vegas, Nevada
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Virginia Health System, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (3):
  - Brussels - UNIV UZ Brussel, Brussels
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (3):
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas
  - Faculdade de Ciencias Medicas da UNICAMP, Campinas
  - Instituto de Oncologia Pediatrica - IOP / GRAAC - UNIFESP, São Paulo
- Canada (4):
  - Kingston General Hospital, Kingston, Ontario
  - CHU Sainte-Justine, Montreal, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzen, Plzen-Lochotin, Plzen - Lochotin
  - University Hospital Motol, Prague
- Rigshospitalet, København, Børneonkologisk Afsnit 5002, Copenhagen, Denmark
- HOP Timone, Marseille, France
- Germany (3):
  - Universitätsklinikum Essen AöR, Essen
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsklinikum Münster, Münster
- University Debrecen Hospital, Debrecen, Hungary
- Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem, Israel
- Italy (4):
  - A.O. Univ. Policlinico "Paolo Giaccone", Palermo
  - Università degli Studi "La Sapienza", Roma
  - Osp. Pediatrico Bambin Gesù, Roma
  - Ospedale Infantile Regina Margherita, Torino
- Children Intensive Care Hosp,Anaesthesiology Dept,Vilnius, Vilnius, Lithuania
- Instituto Nacional de Pediatría, Mexico City, Mexico
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Russia (8):
  - Children Rep.Clin.Hosp of MoH,Cardio Vas.surgery Dept, Kazan, Kazan'
  - Science Res.Instit.CV Diseases,Scientific Res.Dept,Kemerovo, Kemerovo
  - Morozovskaya Children Clin.Hosp.,Haematological Dept, Moscow, Moscow
  - Child.CityClin.Hos.na.ZA Bashlyaeva MoscowHealth Dep,Cardiol, Moscow
  - St.Petersburg State Pediatric Univ.Ministry of Healthcare RF, Saint Petersburg
  - Reg Clin.Hosp.#1,Healthcare Tyumen Region,Cardiovas.Surgery, Tyument
  - State Budget Healthcare Institution "Republican children's clinical hospital", Ufa
  - Childr.CityClin.Hos#9,pediatric&Neonatal Neurol.Ekaterinburg, Yekaterinburg
- Karolinska Univ. sjukhuset, Solna, Sweden
- Universitäts-Kinderspital, Zurich, Switzerland
- Taichung Veterans General Hospital, Taichung, Taiwan
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand
- Turkey (Türkiye) (7):
  - Cukurova Universitesi Tip Fakultesi Cocuk Sagligi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Istanbul Saglik Bilimleri Uni. Kanuni Sultan Suleyman EAH, Istanbul
  - Ege Universitesi Tip Fakultesi Cocuk Hematolojisi Bilim Dali, Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi, Konya
- Ukraine (3):
  - Reg.Children Hosp.Dnipropetrovsk, Dnipropetrovsk
  - Western Ukrainian Spec.Children Med.Center,Lviv, Lviv
  - Reg.Children Hosp,Vinnytsia, Vinnytsia

REFERENCES:
- [Derived] Albisetti M, Tartakovsky I, Halton J, Bomgaars L, Chalmers E, Mitchell LG, Luciani M, Nurmeev I, Gorbatikov K, Miede C, Brueckmann M, Brandao LR; Study Investigators. Dabigatran for Treatment and Secondary Prevention of Venous Thromboembolism in Pediatric Congenital Heart Disease. J Am Heart Assoc. 2024 Feb 20;13(4):e028957. doi: 10.1161/JAHA.122.028957. Epub 2024 Feb 13. PMID 38348778
- [Derived] Brandao LR, Tartakovsky I, Albisetti M, Halton J, Bomgaars L, Chalmers E, Luciani M, Saracco P, Felgenhauer J, Lvova O, Simetzberger M, Sun Z, Mitchell LG. Dabigatran in the treatment and secondary prophylaxis of venous thromboembolism in children with thrombophilia. Blood Adv. 2022 Nov 22;6(22):5908-5923. doi: 10.1182/bloodadvances.2021005681. PMID 36150047
- [Derived] Brandao LR, Albisetti M, Halton J, Bomgaars L, Chalmers E, Mitchell LG, Nurmeev I, Svirin P, Kuhn T, Zapletal O, Tartakovsky I, Simetzberger M, Huang F, Sun Z, Kreuzer J, Gropper S, Brueckmann M, Luciani M; DIVERSITY Study Investigators. Safety of dabigatran etexilate for the secondary prevention of venous thromboembolism in children. Blood. 2020 Feb 13;135(7):491-504. doi: 10.1182/blood.2019000998. PMID 31805182
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open label, single arm prospective cohort study was designed to assess the safety of dabigatran etexilate (DE) for secondary prevention of paediatric venous thromboembolism (VTE) with 12-month (365 days) treatment period followed by 28 days end of treatment follow-up. Results of participants were reported via 3 mutually exclusive age groups.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. 1 enrolled subject was withdrawn before treated due to unable to swallow the capsules.
Groups:
- Dabigatran Etexilate (0 to < 2 Years): Single oral dose of dabigatran etexilate (DE) oral liquid formulation (OLF) ranging from 6.25 milligram(mg) to 143.75 mg was administrated twice daily in the morning and evening for participants aged less than 12 months.
  Single oral dose of DE pellets ranging from 20mg to 330mg was administrated twice daily in the morning and evening for participants aged less than 8 years.
  Dosage of DE was adjusted by age and weight of participants intending to achieve trough plasma dabigatran concentrations between 50 and <250 nanogram(ng)/ milliliter (mL). The DE dose limit was 22.2 mg/kilogram (kg)/day.The maximal DE single dose was 330 mg.
  This arm includes participants aged between 0 to <2 years.
- Dabigatran Etexilate (2 to <12 Years): Single oral dose of DE pellets ranging from 20mg to 330mg was administrated twice daily in the morning and evening for participants aged less than 8 years and who cannot take capsules between 8 and <12 years.
  Single oral dose of DE capsule ranging from 50 mg to 330mg was administrated twice daily in the morning and evening for participants aged at least 8 years.
  Dosage of DE was adjusted by age and weight of participants intending to achieve trough plasma dabigatran concentrations between 50 and <250 ng/mL. The DE dose limit was 22.2 mg/kg/day.The maximal DE single dose was 330 mg.
  This arm includes participants aged between 2 to < 12 years.
- Dabigatran Etexilate (12 to <18 Years): Single oral dose of DE capsule ranging from 50 mg to 330mg was administrated twice daily in the morning and evening for participants aged at least 8 years.
  Dosage of DE was adjusted by age and weight of participants intending to achieve trough plasma dabigatran concentrations between 50 and <250 ng/mL. The DE dose limit was 22.2 mg/kg/day.The maximal DE single dose was 330 mg.
  This arm includes participants aged between 12 to <18 years.
Period: Overall Study
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Started | 9 | 43 | 161
Completed | 8 | 39 | 153
Not Completed | 1 | 4 | 8
Not completed — Other reasons | 0 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all patients who were dispensed trial medication and had taken at least 1 dose of investigational treatment, which was used to assess safety endpoints, demographics and baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years) | Total
Number analyzed (Participants) | 9 | 43 | 161 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 0.6 (0.5) | 6.8 (3.1) | 15.1 (1.6) | 12.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 22 | 70 | 96
  Male | 5 | 21 | 91 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 7 | 9
  Not Hispanic or Latino | 9 | 41 | 153 | 203
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 4 | 8
  White | 8 | 37 | 149 | 194
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Probability of Recurrence of Venous Thromboembolism (VTE) at 6 and 12 Months
Description: The event-free probability of first recurrence of VTE were provided by Kaplan-Meier estimation with its 95% confidence intervals (CIs) at 6 and 12 months.
  Patients who did not experience recurrent VTE at the time of analysis, dropped out from the trial early, were lost to follow-up, or had died from non-VTE related cause were considered as non-events and censored. On treatment period was from first DE administration to 3 days of residual effect period after last DE administration.
Time Frame: At month 6 (Week 26) and 12 (Week 52) of on treatment period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 9 | 43 | 161
Probability
  6 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 0.979 [0.937 to 0.993]
  12 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 0.979 [0.937 to 0.993]

2. Primary Outcome: Event-free Probability of Major or Minor (Including Clinically Relevant Non-major (CRNM)) Bleeding Events at 6 and 12 Months
Description: The event-free probability of major or minor (including CRNM) bleeding event were provided by Kaplan-Meier estimation with its 95% confidence intervals (CIs) at 6 and 12 months.
  Patients who did not experience major or minor (including CRNM) bleeding event at the time of analysis, dropped out from the trial early, were lost to follow-up, or had died from non-bleeding related cause were considered as non-events and censored. On treatment period was from first DE administration to 3 days of residual effect period after last DE administration.
Time Frame: At month 6 (Week 26) and month 12 (Week 52) of on treatment period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 9 | 43 | 161
Probability
  6 months | 0.889 [0.433 to 0.984] | 0.894 [0.706 to 0.965] | 0.753 [0.675 to 0.815]
  12 months | 0.889 [0.433 to 0.984] | 0.831 [0.592 to 0.936] | 0.691 [0.603 to 0.763]

3. Primary Outcome: Event-free Probability of Mortality Overall and Related to Thrombotic or Thromboembolic Events at 6 and 12 Months
Description: The event-free probability of mortality overall and related to thrombotic or thromboembolic events were provided by Kaplan-Meier estimation with its 95% confidence intervals (CIs) at 6 and 12 months.
  Patients who did not experience mortality overall and related to thrombotic or thromboembolic events at the time of analysis, dropped out from the trial early, were lost to follow-up, were considered as non-events and censored. On treatment period was from first DE administration to 3 days of residual effect period after last DE administration.
Time Frame: At month 6 (Week 26) and 12 (Week 52) of on treatment period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 9 | 43 | 161
Probability
  6 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  12 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]

4. Secondary Outcome: Event-free Probability of Occurrence of Post-thrombotic Syndrome (PTS) at 6 and 12 Months
Description: The event-free probability of PTS were provided by Kaplan-Meier estimation with its 95% confidence intervals (CIs) at 6 and 12 months. Patients who did not experience PTS at the time of analysis, dropped out from the trial early, were lost to follow-up, or had died from non-PTS related cause were considered as non-events and censored. On treatment period was from first DE administration to 3 days of residual effect period after last DE administration.
Time Frame: At month 6 (Week 26) and 12 (Week 52) of on treatment period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 9 | 43 | 161
Probability
  6 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 0.979 [0.935 to 0.993]
  12 months | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 0.979 [0.935 to 0.993]

5. Secondary Outcome: Percentage of Participants With Dabigatran Etexilate (DE) Dose Adjustments During on Treatment Period
Description: Percentage of participants with dabigatran etexilate dose adjustments during on treatment period. On treatment period was from first DE administration to 3 days of residual effect period after last DE administration.
Time Frame: From first DE administration to 3 days of residual effect period after last DE administration, up to 52 weeks+ 3 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 9 | 43 | 161
Percentage of participants | 66.7 | 39.5 | 21.1

6. Secondary Outcome: Central Measurement of Activated Partial Thromboplastin Time (aPTT) at Visit 3 (After at Least Six Consecutive Dabigatran Etexilate (DE) Doses)
Time Frame: At Visit 3 (day 4 after first dose of trial medication)
Population: The pharmacodynamics (PD) set (PDS) included all treated patients who provided at least one evaluable PD observation and had no protocol deviations relevant to the evaluation of PD endpoints. Only those with non-missing endpoint values were included in this analysis.
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 8 | 23 | 105
Second (s) | 46.6 (18.1) | 57.1 (70.4) | 56.8 (64.6)

7. Secondary Outcome: Central Measurement of Activated Partial Thromboplastin Time (aPTT) at Post-titration (After at Least 3 Days Following Any Dabigatran Etexilate (DE) Dose Adjustment)
Time Frame: Pharmacodynamics (PD) samples were collected from first dose of trial medication at day 1 and day 4, 22, 43, 85, 127, 183, 239 and 295 until last dose at day 365 and at post-titration (at least 3 days after dose adjustment) if needed, up to 365 days.
Population: The PD set (PDS) included all treated patients who provided at least one evaluable PD observation and had no protocol deviations relevant to the evaluation of PD endpoints. Only those with DE dose adjustment and non-missing endpoint values were included in this analysis.
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 6 | 16 | 31
Second (s) | 49.1 (26.8) | 57.3 (23.9) | 59.0 (80.8)

8. Secondary Outcome: Central Measurement of Ecarin Clotting Time (ECT) at Visit 3 (After at Least Six Consecutive Dabigatran Etexilate (DE) Doses)
Time Frame: At Visit 3 (day 4 after first dose of trial medication)
Population: The pharmacodynamics (PD) set (PDS) included all treated patients who provided at least one evaluable PD observation and had no protocol deviations relevant to the evaluation of PD endpoints. Only those with DE dose adjustment and non-missing endpoint values were included in this analysis.
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 8 | 24 | 105
Second (s) | 52.7 (17.6) | 64.3 (55.7) | 69.5 (30.3)

9. Secondary Outcome: Central Measurement of Ecarin Clotting Time (ECT) at Post-titration (After at Least 3 Days Following Any Dabigatran Etexilate (DE) Dose Adjustment)
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 6 | 16 | 32
Second (s) | 53.3 (19.4) | 66.6 (23.6) | 69.2 (28.7)

10. Secondary Outcome: Central Measurement of Diluted Thrombin Time (dTT) at Visit 3 (After at Least Six Consecutive Dabigatran Etexilate (DE) Doses)
Time Frame: At Visit 3 (day 4 after first dose of trial medication)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 8 | 17 | 64
Second (s) | 37.9 (19.5) | 40.5 (14.6) | 45.3 (17.4)

11. Secondary Outcome: Central Measurement of Diluted Thrombin Time (dTT) at Post-titration (After at Least 3 Days Following Any Dabigatran Etexilate (DE) Dose Adjustment)
Time Frame: dTT values were collected at day 4, 22, 43, 85, 127, 183, 239, and 295 until last dose at day 365 and at post-titration (at least 3 days after dose adjustment) if needed, up to 365 days.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Second (s)
Arm/Group | Dabigatran Etexilate (0 to < 2 Years) | Dabigatran Etexilate (2 to <12 Years) | Dabigatran Etexilate (12 to <18 Years)
Number analyzed (Participants) | 6 | 12 | 26
Second (s) | 40.0 (24.3) | 46.0 (18.6) | 43.4 (17.7)

ADVERSE EVENTS:
Time Frame: From first dose until last dose of study drug + 3 days of residual effect period, up to 52 weeks + 3 days.
Description: The treated set (TS) included all patients who were dispensed trial medication and had taken at least 1 dose of investigational treatment, which was used to assess safety endpoints. The adverse events were reported with single arm align with the study design.
Groups:
- Dabigatran Etexilate (Treated Set): Single oral dose of dabigatran etexilate (DE) oral liquid formulation (OLF) ranging from 6.25 milligram(mg) to 143.75 mg was administrated twice daily in the morning and evening for participants aged less than 12 months.
  Single oral dose of DE pellets ranging from 20mg to 330mg was administrated twice daily in the morning and evening for participants aged less than 8 years.
  Single oral dose of DE capsule ranging from 50 mg to 330mg was administrated twice daily in the morning and evening for participants aged at least 8 years.
  Dosage of DE was adjusted by age and weight of participants intending to achieve trough plasma dabigatran concentrations between 50 and <250 ng/mL. The DE dose limit was 22.2 mg/kg/day.The maximal DE single dose was 330 mg.
Arm/Group | Dabigatran Etexilate (Treated Set)
All-Cause Mortality (participants affected / at risk) | 0/213
Serious Adverse Events (participants affected / at risk) | 30/213
Other Adverse Events (participants affected / at risk) | 113/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Treated Set) (N=213)
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ventricular pre-excitation (Cardiac disorders) | 1
Congenital anomaly (Congenital, familial and genetic disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Hepatic vein stenosis (Hepatobiliary disorders) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pulpitis dental (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Metal poisoning (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ewing's sarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1
Lupus nephritis (Renal and urinary disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bleeding varicose vein (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Lupus vasculitis (Vascular disorders) | 1
Phlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Treated Set) (N=213)
Abdominal pain upper (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 15
Pyrexia (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 34
Upper respiratory tract infection (Infections and infestations) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Headache (Nervous system disorders) | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT02197416/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02197416/SAP_001.pdf